CLINICAL TRIAL: NCT07090460
Title: Pulmonary Overdistension Assessment With Electrical Impedance Tomography in Patients With Acute Respiratory Distress Syndrom in Prone Position.
Acronym: Tomo-BPCO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de la côte Basque (Other)
Responsible Party: Principal Investigator, LABARRERE Séverine, Dr ROZE Hadrien, Centre Hospitalier de la côte Basque
Other Study IDs: P-2025/01; 2025-A00447-42 (Other: ANSM)
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS)
Keywords: Chronic Obstructive Pulmonary Disease; Mechanical Ventilation; NIV; Asynchronies; Electrical Impedance Tomography; Pressure Impedance curve
MeSH Terms: conditions — Respiratory Distress Syndrome; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Mechanical ventilation in COPD requires a good interaction Patient-Ventilator without asynchronies in order to reduce mortality. Dynamic hyperinflation with PEEPi is responsible for major asynchronies in COPD. It is supposed to be symmetrical between the 2 lungs with the same PEEPi. EIT can measure the distribution of tidal ventilation and interlung lung insufflation delay on the impedance time curve of each lung. Moreover, it is possible in intubated COPD patients to assess one lung PEEPi during low flow insufflation with pressure-EIT monitoring.

This study aims to measure interlungs insufflation delay under mechanical ventilation in COPD patients

DETAILED DESCRIPTION:
Scientific justification: Moderate or severe COPD with respiratory acidosis requires mechanical ventilation whether it is non-invasive or after intubation. There is a risk of various asynchronies due to dynamic hyperinflation, and it has been shown that a high level of asynchronies can be associated with mortality. EIT can measure the regional distribution of tidal ventilation, and its timing. It can also measure unilateral Pressure-EIT curves with low inflection point representing PEEPi.

Strategy description: Patients with moderate or severe COPD treated with mechanical ventilation equipped with EIT will be included. EIT will be monitored during tidal ventilation and during PEEP titration by the attending physician as it is already done in our unit. In case of invasive ventilation (NIV failure), a classical low flow PV curve will be done in order to mesure one lung PEEPi. For that the acquisition of EIT data during the low flow PV curve will be analysed secondary with a dedicated software. Reconstruction of EIT derived PV curve will determine the regional PEEPi.

Follow up description:

* Measurement of EIT data and ventilator spirometry during NIV initiation and PEEP titration.
* Blood gases under NIV as usual
* Hemodynamic data

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the ICU and who suffered moderate or severe COP (Gold 3 and 4)), with respiratory acidosis under NIV or intubated, and equipped with EIT over the age of 18.

Exclusion Criteria:

* Broncho-pleural leaks
* Pregnant or breastfeeding woman.
* Guardianship or curatorship
* Deprived of liberty
* No health insurance
* Impossibility to correctly position the EIT belt (e.g., dressings, chest drainage, etc.)
* Contra indications to EIT (e.g., implantable cardiac defibrillator, pacemaker, instable spinal lesions)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Respiratory Distress Syndrom in prone position
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Assessing inter-lungs insufflation delay under NIV or invasive mechanical ventilation on the impedance-time curves without PEEP. | Only 1 visit

SECONDARY OUTCOMES:
Assessing inter-lungs insufflation delay under NIV or invasive mechanical ventilation on the impedance-time curves with PEEP. | Only 1 visit
Comparison of End Expiratory Lung Impedance with or without PEEP | Only 1 visit
Post treatment analysis of EIT low flow PV curves in intubated sedated patients, measurement of each lung PEEPi | Only 1 visit

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Côte Basque, Bayonne, Centre Hospitalier de La Côte Basque, France

IPD SHARING:
Plan to Share IPD: No